CLINICAL TRIAL: NCT02301546
Title: Cognitive Training and Practice Effects in Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kevin Duff, Associate Professor of Neurology, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01AG045163 (NIH); R01AG045163 (NIH)
Record Dates: First submitted 2014-11-21; First posted 2014-11-26 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- experimental cognitive training (Experimental): Participants will use experimental computerized cognitive training exercises, 1 hour per day, 3 - 5 days per week, for 13 weeks.
  Interventions: Behavioral: computerized cognitive exercises
- control cognitive exercises (Active Comparator): Participants will use control computerized cognitive activities, 1 hour per day, 3 - 5 days per week, for 13 weeks.
  Interventions: Behavioral: computerized cognitive exercises

INTERVENTIONS:
Behavioral: computerized cognitive exercises — Each group will perform computerized cognitive exercises, 1 hour per day, 3 - 5 days per week, for 13 weeks. The experimental group will use exercises shown to improve cognition, whereas the comparator group will use exercises without clear beneficial findings.

SUMMARY:
The current study will test the effectiveness of a computerized cognitive training program on auditory memory and attention in patients with mild cognitive impairment. Practice effects will also be examined as a moderator of treatment response.

DETAILED DESCRIPTION:
The current study will test the effectiveness of a computerized cognitive (thinking) training program on improving thinking and memory in patients with mild cognitive impairment. The investigators will also examine how short term changes in thinking abilities (i.e., practice effects) can be related to improvement in thinking abilities after the cognitive training program.

ELIGIBILITY:
Inclusion Criteria:

* Mild Cognitive Impairment, amnestic subtype

  * 65 years of age or older
  * Availability of a knowledgeable informant
* Access to internet 3 hours per week
* Adequate vision, hearing, and motor responding to participate in training

Exclusion Criteria:

* History of major stroke, head injury with loss of consciousness of >30 minutes, or other neurological disorder or systemic illness that are thought to be affecting cognition (e.g., seizure disorder, demyelinating disorder, etc.)
* Current or past major psychiatric illness (e.g., schizophrenia, bipolar affective disorder)
* History of substance abuse
* Current use of antipsychotics or anticonvulsant medications
* Currently residing in a nursing home or other skilled nursing facility

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 197 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Duff, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Center for Alzheimer's Care, Imaging and Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Other researchers can contact the PI to request copies of the study data.

REFERENCES:
- [Derived] Duff K, Ying J, Suhrie KR, Dalley BCA, Atkinson TJ, Porter SM, Dixon AM, Hammers DB, Wolinsky FD. Computerized Cognitive Training in Amnestic Mild Cognitive Impairment: A Randomized Clinical Trial. J Geriatr Psychiatry Neurol. 2022 May;35(3):400-409. doi: 10.1177/08919887211006472. Epub 2021 Mar 30. PMID 33783254

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 51 individuals were enrolled in the study but were withdrawn by the research team because they did not meet criteria for amnestic Mild Cognitive Impairment on objective testing.
Period: Short-term Effectiveness (~13 Weeks)
Arm/Group | Experimental Cognitive Training | Control Cognitive Exercises
Started | 73 | 73
Completed | 55 | 58
Not Completed | 18 | 15
Not completed — Withdrawal by Subject | 7 | 8
Not completed — non-compliant | 10 | 7
Not completed — screen fail | 1 | 0
Period: Long Term Effectiveness (~1 Year)
Arm/Group | Experimental Cognitive Training | Control Cognitive Exercises
Started | 55 | 58
Completed | 43 | 51
Not Completed | 12 | 7
Not completed — Lost to Follow-up | 3 | 3
Not completed — Death | 2 | 0
Not completed — Withdrawal by Subject | 6 | 2
Not completed — moved away | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Cognitive Training | Control Cognitive Exercises | Total
Number analyzed (Participants) | 55 | 58 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.9 (6.3) | 75.0 (5.8) | 75.0 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 29 | 33 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 54 | 57 | 111
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 55 | 58 | 113
one week practice effects [Mean (Standard Deviation); unit: z-score units] — This measure indicates how much a participant improves from baseline to one week on a composite of seven cognitive scores (i.e., practice effects). The practice effects on the seven cognitive scores are averaged to get the composite. The presented value is a z-score, which has a theoretical mean of 0 and a standard deviation of +/-1. Expected range should be approximately -4 to +4. Higher scores indicate better than expected practice effects compared to normative data. Participants are not assigned to an intervention until after this one week score is collected. This is not an outcome measure.
  z-score units | -0.4 (0.7) | -0.4 (0.7) | -0.4 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Auditory Memory Attention Index
Description: This is a composite of six subtests of the Repeatable Battery for the Assessment of Neuropsychological Status. It is a standard score (mean=100, standard deviation=15), with a range of approximately 45 - 145, with higher scores indicating better outcome.
Time Frame: 13 weeks
Population: Mixed effects model
Measure: Mean (Standard Deviation); unit: standard score units
Arm/Group | Experimental Cognitive Training | Control Cognitive Exercises
Number analyzed (Participants) | 55 | 58
standard score units | 89.0 (13.1) | 94.3 (12.1)
Statistical Analysis 1: Comparison: Experimental Cognitive Training vs Control Cognitive Exercises; Test type: Superiority; p < 0.01, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: approximately 13 weeks
Arm/Group | Experimental Cognitive Training | Control Cognitive Exercises
All-Cause Mortality (participants affected / at risk) | 2/73 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/73
Other Adverse Events (participants affected / at risk) | 0/73 | 0/73

LIMITATIONS AND CAVEATS:
underpowered

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT02301546/Prot_SAP_000.pdf